CLINICAL TRIAL: NCT06752863
Title: Comparative Study of Labetalol Infusion Versus Dexmedetomidine Infusion in Hypotensive Anesthesia in Ear, Nose and Throat Surgeries
Brief Title: Labetalol Infusion and Dexmedetomidine Infusion in Hypotensive Anesthesia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU MD105/2024
Record Dates: First submitted 2024-12-21; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-06

CONDITIONS: Hypotensive Anesthesia; Ear, Nose and Throat Procedure
Keywords: Hypotensive anesthesia; Labetalol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Masking Description: data collector is also masked in the clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients undergoing ear, nose and throat surgeries who will receive dexmedetomidine infusion (Active Comparator): Dexmedetomidine group: the patients will receive deliberate hypotensive anesthesia with dexmedetomidine infusion (precedex ® 200 μg/2 ml; Hospira, Inc., Rocky Mount, USA) via syringe pump by adding 200 mcg (2ml) of dexmedetomidine to 48 ml of normal saline (final concentration of 4 mcg/ml) The patients will receive a loading dose of 1mcg/kg intravenously followed by an infusion of 0.7 mcg/kg/hour as maintenance dose.
  Interventions: Drug: Hypotensive anesthesia in ear, nose and throat surgeries using labetalol and dexmedetomidine infusions
- Patients undergoing ear, nose and throat surgeries who will receive Labetalol infusion (Active Comparator): Labetalol groups: the patients will receive deliberate hypotensive anesthesia with labetalol infusion (Labipress 100mg/20ml; Al Debeiky pharma(DBK) pharmaceutical co., Cairo, Egypt) via syringe pump by adding 100 mg (20ml) of Labetalol to 30ml of normal saline (final concentration of 2 mg/ml) The patients will receive a loading dose of 0.4mg/kg intravenously followed by an infusion of 0.04mg/kg/hour as maintenance dose.
  Interventions: Drug: Hypotensive anesthesia in ear, nose and throat surgeries using labetalol and dexmedetomidine infusions

INTERVENTIONS:
Drug: Hypotensive anesthesia in ear, nose and throat surgeries using labetalol and dexmedetomidine infusions — The study compares the role of Labetalol infusion versus Dexmedetomidine infusion in hypotensive anesthesia in patients having ear, nose and throat surgeries

SUMMARY:
this study aims to compare between the role of Labetalol infusion versus Dexmedetomidine infusion in hypotensive anesthesia in Ear, Nose and Throat surgeries.

DETAILED DESCRIPTION:
Hypotensive anaesthesia is the deliberate lowering of a patient's blood pressure during surgery. It is necessary during ear, nose and throat surgery for drying surgical field, ease in operation procedure and shortening of the duration of surgery. Labetalol is a unique parenteral anti-hypertensive drug that has selective α1 and non- selective β adrenergic antagonist effects. In humans, the β to α blocking potency ratio is 7: 1 for IV labetalol. Dexmedetomidine is highly selective alpha2 adrenergic agonist having several beneficial actions during the perioperative period. Activation of alpha2 adrenergic receptors in the brain and spinal cord inhibits neuronal firing causing hypotension and bradycardia. This study was designed to compare between the role of Labetalol infusion versus Dexmedetomidine infusion in hypotensive anesthesia in Ear, Nose and Throat surgeries.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists I, II (ASA I, II) patients who were candidate for Ear, Nose and Throat surgeries.
* Age: between 20 and 50 years

Exclusion Criteria:

* Patients with uncontrolled hypertension, variable degrees of heart block, congestive cardiac failure, coagulopathy, cerebral insufficiency, hepatic or renal abnormality
* Patients on beta blocker or clonidine
* Pregnant or lactating females
* Patients who were allergic to any of the anesthetic or hypotensive drugs used in the study
* Patient refusal to be included in the trial

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean arterial blood pressure changes before induction of anesthesia & every 15 min throughout deliberate hypotension | 12 months

SECONDARY OUTCOMES:
Heart rate changes before induction of anesthesia and every 15 min | 12 months
Surgical site oligaemia will be evaluated by the surgeons by rating the amount of bleeding according to Modena bleeding score that provides five different levels (from "Grade 1 - no bleeding" to "Grade 5") | 12 months
Surgeon satisfaction At the end of the surgery will be evaluated by one surgeon and recorded according to a 5-point Likert scale (5: excellent, 4: Good, 3: Satisfactory, 2: Poor, 1: Very poor) | 12 months
Total anesthetic consumption including both inhalational anesthetic consumption and narcotics consumption. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided